CLINICAL TRIAL: NCT00675948
Title: An Open-label, Extension Study, to Investigate the Long-term Safety and Tolerability of Cannabis Based Medicine Extracts in Patients With Cancer-related Pain.
Brief Title: Study to Compare the Safety and Tolerability of Sativex® in Patients With Cancer Related Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GWEXT0101
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pain; Cancer
Keywords: Palliative Care; Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental): Active treatment
  Interventions: Drug: Sativex
- GW-2000-02 (Experimental): Active treatment
  Interventions: Drug: GW-2000-02

INTERVENTIONS:
Drug: Sativex — Containing delta-9-tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml; both as extract of Cannabis sativa L.
  Subjects received study medication delivered in 100 µl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three hour period and 48 actuations (THC 130 mg:CBD 120 mg) in 24 hours.
  Other Names: GW-1000-02
  Arms: Sativex
Drug: GW-2000-02 — Containing THC, 27 mg/ml, as extract of Cannabis sativa L. Subjects received study medication delivered in 100 µl actuations by a pump action oromucosal spray. Maximum permitted dose was eight actuations in any three hour period and 48 actuations (THC 130 mg) in 24 hours.
  Arms: GW-2000-02

SUMMARY:
The purpose of this study is to assess the safety and tolerability of long term therapy with Sativex® and GW-2000-02.

DETAILED DESCRIPTION:
Subjects who have previously participated in GWCA0101, a two week (two days baseline and two weeks treatment period), multicentre, double blind, randomised, placebo controlled, parallel group study to evaluate the efficacy of Sativex® (containing delta-9-tetrahydrocannabinol [THC] and cannabidiol [CBD]) and GW-2000-02 (containing THC alone) in subjects with cancer-related pain are screened, and if eligible begin dosing with open-label Sativex®. They are allowed to self-titrate their study medication to symptom resolution or maximum tolerated/allowable dose of 130 mg THC and 120 mg CBD and have the opportunity to request a change from Sativex® to GW-2000-02 if they or the investigator consider their response less than optimal. Subjects are reviewed for tolerability and evidence of clinical benefit at 7-10 days after Visit 1 and then every four weeks. Continuation within the study is conditional on satisfactory reports of tolerability, efficacy and dosing regime.

ELIGIBILITY:
Inclusion Criteria:

* Willing and eligible to continue into the extension study from GWCA0101.
* Complied adequately with the study requirements, as detailed in GWCA0101.
* In the investigator's opinion able to undertake and comply with all of the study requirements (it is understood that progress of the disease may accelerate and affect this ability).
* Willing and able to read, consider and understand the subject information and consent form and to give written informed consent in compliance with the Declaration of Helsinki1.
* Willing to allow their own general practitioner, and consultant if appropriate, to be informed of study participation.
* Willing for their name to be notified to the Home Office for participation in the trial.

Exclusion Criteria:

* Have not participated in GWCA0101.
* Have not complied adequately with the study requirements, as detailed in GWCA0101.
* Experienced an unacceptable adverse event, whilst participating in GWCA0101.
* Known or suspected to have had an adverse reaction to cannabinoids causing psychosis or other severe psychiatric illness.
* History of any type of schizophrenia, any other psychotic illness, a serious personality disorder, or other significant psychiatric illness other than depression associated with their chronic pain and/or in response to the underlying condition.
* Currently taking levodopa (Sinemet®, Sinemet plus®, Levodopa®, L-dopa®, Madopar®, Benserazide®).
* Has a serious cardiovascular disorder, including angina, uncontrolled hypertension, or an uncontrolled symptomatic cardiac arrhythmia.
* Has significant renal or hepatic impairment, which in the opinion of the investigator, are unsuitable for treatment with Investigational Medicinal Product.
* History of epilepsy.
* Female subjects of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.
* If female, are pregnant or lactating, or are planning pregnancy during the course of the study and for three months thereafter.
* Have oral cavity cancers or whose previous treatments had included radiotherapy to the floor of the mouth.
* In the opinion of the investigator, are unsuitable to participate in the study for any other reason, not mentioned in the inclusion and exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy R Johnson, MB ChB, Principal Investigator — Shropshire and Mid-Wales Hospice
Locations (1):
- Shropshire and Mid-Wales Hospice, Shrewsbury, United Kingdom

REFERENCES:
- [Result] Johnson JR, Lossignol D, Burnell-Nugent M, Fallon MT. An open-label extension study to investigate the long-term safety and tolerability of THC/CBD oromucosal spray and oromucosal THC spray in patients with terminal cancer-related pain refractory to strong opioid analgesics. J Pain Symptom Manage. 2013 Aug;46(2):207-18. doi: 10.1016/j.jpainsymman.2012.07.014. Epub 2012 Nov 8. PMID 23141881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was recruited on the 30th April 2002
Groups:
- Sativex: Each 100 μl actuation of Sativex delivered a dose containing 2.7 mg THC and 2.5 mg CBD
- THC Alone: Each 100 μl actuation of THC alone delivered a dose containing 2.7 mg THC
Period: Overall Study
Arm/Group | Sativex | THC Alone
Started | 39 | 4
Completed | 0 | 1
Not Completed | 39 | 3
Not completed — Adverse Event | 23 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Pain under control | 1 | 0
Not completed — Sponsor decision | 0 | 1
Not completed — Patient died | 1 | 0
Not completed — Patient unable to comply with diaries | 1 | 0
Not completed — Patient feels unable to take medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | THC Alone | Total
Number analyzed (Participants) | 39 | 4 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 4 | 33
  >=65 years | 10 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.5) | 58.6 (6.28) | 57.6 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 19
  Male | 23 | 1 | 24
Region of Enrollment [Number; unit: participants]
  United Kingdom | 31 | 3 | 34
  Belgium | 8 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Adverse Events as a Measure of Subject Safety
Description: The number of subjects who experienced an adverse event in this study is presented.
Time Frame: 0 - 657 days
Population: All subjects who took at least one dose of study medication and yielded on-treatment efficacy data were classed as the safety population.
Measure: Number; unit: participants
Groups:
- Sativex: Each 100 μl actuation of Sativex delivered a dose containing 2.7 mg delta-9-tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD)
Arm/Group | Sativex | THC Alone
Number analyzed (Participants) | 39 | 4
participants | 37 | 4

2. Secondary Outcome: Change From Baseline in the Mean Brief Pain Inventory (Short Form) - Pain Severity Score at the End of Treatment
Description: The Brief Pain Inventory (Short Form) is a 14-item questionnaire that asks subjects to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The severity composite score was calculated as the arithmetic mean of the four severity items (range 0-10). The minimum value is zero and maximum is 10. A negative value indicates an improvement in score from baseline. The end of treatment was classed as study completion or withdrawal, if this occurred sooner. Calculation of the mean Brief Pain Inventory (Short Form) score was only carried out when data was available for 10 or more subjects at the relevant study visits. As such, no mean scores were calculated for subjects taking THC alone.
Time Frame: 0 - 657 days
Population: The efficacy analyses were conducted on data from all subjects who entered the study, who were randomised, who received at least one dose of study medication and who yielded on-treatment efficacy data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone
Number analyzed (Participants) | 17 | 0
units on a scale | -0.53 (1.28) |

3. Secondary Outcome: Change From Baseline in the Mean EORTC Quality of Life-C30 Questionnaire - Global Health Status Score at the End of Treatment
Description: The EORTC Quality of Life-C30 Health Status visual analogue scale was a self-reported score where subjects rated their health state from: 0 = worst health state imaginable to 100 = best health state imaginable. An increase in score from baseline indicates an improvement in condition. The end of treatment was classed as study completion or withdrawal, if this occurred sooner. Calculation of mean EORTC Quality of Life-C30 Health Status scores was only produced when data was available for 10 or more subjects at the relevant study visits. As such, no mean scores were calculated for subjects taking THC alone.
Time Frame: 0 - 657 days
Population: The efficacy analyses were conducted on data from all randomised subjects who received at least one dose of study medication and who yielded on-treatment efficacy data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | THC Alone
Number analyzed (Participants) | 17 | 0
units on a scale | -2.0 (28.34) |

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring from the time of consent to post study follow up (2 - 521 days) were collected. All deaths and serious adverse events (SAEs) occurring within 28 days of the final dose of study medication were also collected.
Description: All AEs occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | THC Alone
Serious Adverse Events (participants affected / at risk) | 20/39 | 1/4
Other Adverse Events (participants affected / at risk) | 37/39 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=39) | THC Alone (N=4)
Anaemia NOS aggravated (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction NOS (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Weakness (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis NOS (Infections and infestations) | 1 | 0
Sepsis NOS (Infections and infestations) | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 1 | 0
Accident NOS (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 1
Metastases to brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuropathic pain (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Renal Failure NOS (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=39) | THC Alone (N=4)
Nausea (Gastrointestinal disorders) | 10 | 0
Vomiting (Gastrointestinal disorders) | 10 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dizziness (Nervous system disorders) | 8 | 1
Somnolence (Nervous system disorders) | 8 | 0
Headache (Nervous system disorders) | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 7 | 1
Pain in limb (Musculoskeletal and connective tissue disorders) | 8 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastritis NOS (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Thirst (General disorders) | 2 | 0
Weakness (General disorders) | 2 | 0
Lower respiratory tract infection NOS (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Liver function tests abnormal (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Pain in back (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 1
Metastasis to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Jerky movement (Nervous system disorders) | 2 | 0
Clonic convulsions (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Disorientation (Psychiatric disorders) | 2 | 0
Hallucination NOS (Psychiatric disorders) | 2 | 0
Affect lability (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 3 | 0
Renal failure NOS (Renal and urinary disorders) | 0 | 1
Renal Impairment NOS (Renal and urinary disorders) | 0 | 1
Rash NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion NOS (Vascular disorders) | 0 | 1
Hypotension NOS (Vascular disorders) | 2 | 0
Hot flushes NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Policy:

GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications for example, manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.